CLINICAL TRIAL: NCT00586664
Title: Efficacy and Safety Study of Bepotastine Besilate Ophthalmic Solution in Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-S&E-0409071-P
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine besilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% (Experimental)
  Interventions: Drug: Bepreve (bepotastine besilate ophthalmic solution) 1.5%
- Bepotastine Besilate Ophthalmic Solution 1.0% (Experimental)
  Interventions: Drug: Bepotastine Besilate Ophthalmic Solution 1.0%
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: Bepreve (bepotastine besilate ophthalmic solution) 1.5% — sterile ophthalmic solution
  Arms: Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5%
Drug: placebo comparator — sterile ophthalmic solution
  Arms: Placebo
Drug: Bepotastine Besilate Ophthalmic Solution 1.0% — sterile ophthalmic solution
  Arms: Bepotastine Besilate Ophthalmic Solution 1.0%

SUMMARY:
Efficacy and safety study of bepotastine besilate ophthalmic solution in allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 10 years of age

Exclusion Criteria:

* No active ocular disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

REFERENCES:
- [Derived] Meier EJ, Torkildsen GL, Gow JA, McNamara TR, Gomes PJ, Williams JI; Bepotastine Besilate Ophthalmic Solutions Study Group. Integrated phase III trials of bepotastine besilate ophthalmic solution 1.5% for ocular itching associated with allergic conjunctivitis. Allergy Asthma Proc. 2012 May-Jun;33(3):265-74. doi: 10.2500/aap.2012.33.3570. PMID 22991696
- [Derived] Macejko TT, Bergmann MT, Williams JI, Gow JA, Gomes PJ, McNamara TR, Abelson MB; Bepotastine Besilate Ophthalmic Solutions Clinical Study Group. Multicenter clinical evaluation of bepotastine besilate ophthalmic solutions 1.0% and 1.5% to treat allergic conjunctivitis. Am J Ophthalmol. 2010 Jul;150(1):122-127.e5. doi: 10.1016/j.ajo.2010.02.007. Epub 2010 May 20. PMID 20488431

RESULTS

PARTICIPANT FLOW:
Groups:
- Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5%; Placebo; Bepotastine Besilate Ophthalmic Solution 1.0%: 1 drop, both eyes at 3 different time points post-CAC within 3 different time points post-dose, for a total of 9 separate time points
Period: Overall Study
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Started | 43 | 43 | 44
Completed | 38 | 36 | 43
Not Completed | 5 | 7 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 1
Not completed — Exclusion criteria met | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0% | Total
Number analyzed (Participants) | 43 | 43 | 44 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 33.3 (15.1) | 33.3 (14.1) | 34.8 (14.0) | 33.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 25 | 75
  Male | 22 | 14 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular Itching score: 0=None; 0.5=Intermittent tickle sensation possibly localized in the corner of the eye; 1.0=Intermittent tickle sensation involving more than the corner of the eye; 1.5=Intermittent all-over tickling sensation; 2.0=Mild continuous itch (can be localized) without desire to rub; 2.5=Moderate, diffuse continuous itch with desire to rub; 3.0=Severe itch with desire to rub; 3.5=Severe itch improved with minimal rubbing; 4.0=Incapacitating itch with irresistible urge to rub
Time Frame: 15 minutes, 8 hours & 16 hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 3 minute post CAC | 0.4 (0.6) | 1.9 (1.0) | 0.4 (0.7)
  15 Minutes post-dose: 5 minute post CAC | 0.5 (0.6) | 2.1 (1.1) | 0.6 (0.7)
  15 Minutes post-dose: 7 minute post CAC | 0.5 (0.6) | 1.9 (1.2) | 0.6 (0.7)
  8 Hours post-dose: 3 minute post CAC | 0.9 (0.9) | 2.2 (1.0) | 1.0 (0.8)
  8 Hours post-dose: 5 minute post CAC | 1.0 (0.8) | 2.3 (1.1) | 1.0 (0.7)
  8 Hours post-dose: 7 minute post CAC | 0.9 (0.8) | 2.1 (1.1) | 0.9 (0.7)
  16 Hours post-dose: 3 minute post CAC | 1.2 (0.8) | 1.8 (1.0) | 1.3 (0.8)
  16 Hours post-dose: 5 minute post CAC | 1.4 (1.0) | 2.2 (1.1) | 1.4 (0.8)
  16 Hours post-dose: 7 minute post CAC | 1.2 (0.9) | 2.0 (1.0) | 1.2 (0.8)

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 minutes, 8 hours & 16 hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 minute post CAC | 1.4 (0.7) | 1.9 (0.6) | 1.3 (0.7)
  15 Minutes post-dose: 15 minute post CAC | 1.6 (0.8) | 2.0 (0.6) | 1.5 (0.8)
  15 Minutes post-dose: 20 minute post CAC | 1.7 (0.8) | 1.9 (0.7) | 1.6 (0.7)
  8 Hours post-dose: 7 minute post CAC | 1.3 (0.7) | 1.7 (0.7) | 1.3 (0.7)
  8 Hours post-dose: 15 minute post CAC | 1.5 (0.8) | 1.9 (0.6) | 1.6 (0.6)
  8 Hours post-dose: 20 minute post CAC | 1.6 (0.8) | 1.9 (0.7) | 1.6 (0.7)
  16 Hours post-dose: 7 minute post CAC | 1.8 (0.7) | 1.9 (0.6) | 1.5 (0.8)
  16 Hours post-dose: 15 minute post CAC | 1.9 (0.9) | 2.0 (0.7) | 1.6 (0.8)
  16 Hours post-dose: 20 minute post CAC | 1.9 (0.8) | 2.0 (0.7) | 1.6 (0.9)

3. Secondary Outcome: Ciliary Redness
Description: Ciliary Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minute post CAC | 1.4 (0.7) | 1.9 (0.7) | 1.2 (0.7)
  15 Minutes post-dose: 15 Minute post CAC | 1.7 (0.7) | 2.1 (0.7) | 1.5 (0.8)
  15 Minutes post-dose: 20 Minute post CAC | 1.7 (0.8) | 1.9 (0.8) | 1.6 (0.8)
  8 Hours post-dose: 7 Minute post CAC | 1.6 (0.8) | 1.8 (0.6) | 1.3 (0.7)
  8 Hours post-dose: 15 Minute post CAC | 1.8 (0.7) | 2.0 (0.7) | 1.6 (0.8)
  8 Hours post-dose: 20 Minute post CAC | 1.8 (0.7) | 1.9 (0.7) | 1.6 (0.8)
  16 Hours post-dose: 7 Minute post CAC | 1.7 (0.9) | 1.9 (0.8) | 1.4 (0.8)
  16 Hours post-dose: 15 Minute post CAC | 1.9 (0.9) | 2.1 (0.8) | 1.7 (0.9)
  16 Hours post-dose: 20 Minute post CAC | 1.9 (0.9) | 2.1 (0.9) | 1.7 (0.9)

4. Secondary Outcome: Episcleral Redness
Description: Episcleral Redness score: 0=None; 1.0=Mild-Slightly dilated blood vessels; color of vessels typically pink; 2.0=Moderate-More apparent dilation of blood vessels; vessel color more intense (redder); 3.0=Severe-Numerous, obvious dilated blood vessels; absence of chemosis color is deep red, presence of chemosis may be less red or pink; 4.0=Extremely severe-Large, numerous dilated blood vessels characterized by severe deep red color regardless of chemosis grade
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minute post-dose: 7 Minutes post CAC | 1.5 (0.8) | 2.0 (0.6) | 1.3 (0.7)
  15 Minute post-dose: 15 Minutes post CAC | 1.7 (0.8) | 2.1 (0.7) | 1.6 (0.8)
  15 Minute post-dose: 20 Minutes post CAC | 1.8 (0.8) | 2.0 (0.8) | 1.9 (0.8)
  8 Hours post-dose: 7 Minutes post CAC | 1.7 (0.8) | 2.0 (0.6) | 1.5 (0.8)
  8 Hours post-dose: 15 Minutes post CAC | 1.9 (0.8) | 2.1 (0.7) | 1.7 (0.8)
  8 Hours post-dose: 20 Minutes post CAC | 2.0 (0.7) | 2.0 (0.7) | 1.7 (0.9)
  16 Hours post-dose: 7 Minutes post CAC | 1.8 (0.9) | 2.0 (0.7) | 1.5 (0.9)
  16 Hours post-dose: 15 Minutes post CAC | 1.9 (0.9) | 2.2 (0.8) | 1.8 (0.9)
  16 Hours post-dose: 20 Minutes post CAC | 2.0 (0.9) | 2.1 (0.9) | 1.8 (1.0)

5. Secondary Outcome: Chemosis
Description: Chemosis score: 0 = None; 1.0 = Mild-Detectable only by slit lamp beam; definite separation of conjunctiva from sclera; 2.0 = Moderate-Visible in normal room light; more diffuse edema; 3.0 = Severe-Conjunctival billowing at the limbus; very diffuse and noticeable; 4.0 = Extremely severe-Overall ballooning of conjunctiva
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.3 (0.5) | 0.5 (0.7) | 0.3 (0.4)
  15 Minutes post-dose: 15 Minutes post CAC | 0.4 (0.5) | 0.7 (0.8) | 0.3 (0.5)
  15 Minutes post-dose: 20 Minutes post CAC | 0.4 (0.5) | 0.7 (0.8) | 0.4 (0.5)
  8 Hours post-dose: 7 Minutes post CAC | 0.5 (0.5) | 0.6 (0.7) | 0.4 (0.6)
  8 Hours post-dose: 15 Minutes post CAC | 0.5 (0.6) | 0.8 (0.8) | 0.5 (0.7)
  8 Hours post-dose: 20 Minutes post CAC | 0.5 (0.7) | 0.8 (0.8) | 0.6 (0.8)
  16 Hours post-dose: 7 Minutes post CAC | 0.5 (0.5) | 0.5 (0.6) | 0.4 (0.6)
  16 Hours post-dose: 15 Minutes post CAC | 0.5 (0.6) | 0.8 (0.7) | 0.6 (0.8)
  16 Hours post-dose: 20 Minutes post CAC | 0.6 (0.6) | 0.8 (0.7) | 0.6 (0.9)

6. Secondary Outcome: Eyelid Swelling
Description: Eyelid Swelling score: 0 = None; 1.0 = Mild-Detectable swelling of lower and/or upper lid; 2.0 = Moderate-Definite swelling of lower and/or upper lid; 3.0 = Severe-Swelling of lower and/or upper lid to the point that there is a decrease in the space between your upper and lower lids
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.2 (0.4) | 0.5 (0.8) | 0.2 (0.3)
  15 Minutes post-dose: 15 Minutes post CAC | 0.3 (0.5) | 0.5 (0.7) | 0.2 (0.4)
  15 Minutes post-dose: 20 Minutes post CAC | 0.3 (0.6) | 0.5 (0.7) | 0.3 (0.5)
  8 Hours post-dose: 7 Minutes post CAC | 0.2 (0.4) | 0.6 (0.8) | 0.2 (0.4)
  8 Hours post-dose: 15 Minutes post CAC | 0.3 (0.5) | 0.7 (0.8) | 0.3 (0.7)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.5) | 0.6 (0.8) | 0.4 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 0.3 (0.5) | 0.6 (0.7) | 0.2 (0.4)
  16 Hours post-dose: 15 Minutes post CAC | 0.3 (0.6) | 0.8 (0.8) | 0.2 (0.4)
  16 Hours post-dose: 20 Minutes post CAC | 0.4 (0.5) | 0.6 (0.7) | 0.3 (0.5)

7. Secondary Outcome: Rhinorrhea (Runny Nose)
Description: Rhinorrhea score: 0 = None; 1.0 = Mild-Sensation of nasal mucus flowing down nasal passage; no discharge present; 2.0 = Moderate-May be associated with post-nasal drip; nasal mucus flow more pronounced; will need to blow nose soon; 3.0 = Moderate/Severe-Nasal mucus discharge requiring occasional wiping with Kleenex; 4.0 = Severe-Uncontrolled nasal discharge; requiring frequent wiping and blowing nose
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.2 (0.6) | 0.9 (1.0) | 0.3 (0.5)
  15 Minutes post-dose: 15 Minutes post CAC | 0.3 (0.7) | 1.1 (1.1) | 0.3 (0.6)
  15 Minutes post-dose: 20 Minutes post CAC | 0.3 (0.7) | 0.7 (0.8) | 0.3 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.3 (0.7) | 1.0 (1.1) | 0.3 (0.6)
  8 Hours post-dose: 15 Minutes post CAC | 0.2 (0.6) | 1.2 (1.2) | 0.5 (0.8)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.5) | 0.9 (1.0) | 0.5 (0.9)
  16 Hours post-dose: 7 Minutes post CAC | 0.7 (0.9) | 1.0 (1.2) | 0.7 (0.8)
  16 Hours post-dose: 15 Minutes post CAC | 0.6 (0.8) | 1.3 (1.3) | 0.7 (0.8)
  16 Hours post-dose: 20 Minutes post CAC | 0.6 (0.9) | 1.1 (1.2) | 0.7 (0.8)

8. Secondary Outcome: Nasal Pruritus (Itchy Nose)
Description: Nasal Pruritus score: 0 = None; 1.0 = Mild-An intermittent tickle sensation; 2.0 = Moderate-A mild continuous itch; 3.0 = Moderate/Severe-A severe itch with desire to rub; 4.0 = Severe-Incapacitating itch with an irresistible urge to rub
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.1 (0.4) | 0.4 (0.8) | 0.1 (0.3)
  15 Minutes post-dose: 15 Minutes post CAC | 0.2 (0.6) | 0.4 (0.8) | 0.2 (0.5)
  15 Minutes post-dose: 20 Minutes post CAC | 0.2 (0.5) | 0.5 (0.9) | 0.2 (0.6)
  8 Hours post-dose: 7 Minutes post CAC | 0.1 (0.5) | 0.5 (0.8) | 0.2 (0.5)
  8 Hours post-dose: 15 Minutes post CAC | 0.2 (0.7) | 0.6 (1.0) | 0.3 (0.6)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.7) | 0.6 (1.0) | 0.4 (0.7)
  16 Hours post-dose: 7 Minutes post CAC | 0.3 (0.6) | 0.6 (1.1) | 0.3 (0.5)
  16 Hours post-dose: 15 Minutes post CAC | 0.3 (0.6) | 0.7 (0.9) | 0.5 (0.7)
  16 Hours post-dose: 20 Minutes post CAC | 0.3 (0.7) | 0.7 (1.0) | 0.5 (0.8)

9. Secondary Outcome: Ear or Palate Pruritus (Itchy Ear or Palate)
Description: Ear or Palate Pruritus score: 0 = None; 1.0 = Mild-An intermittent tickle sensation; 2.0 = Moderate-A mild continuous itch; 3.0 = Moderate/Severe-A severe itch with desire to rub; 4.0 = Severe-Incapacitating itch with an irresistible urge to rub
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.1 (0.3) | 0.3 (0.5) | 0.2 (0.4)
  15 Minutes post-dose: 15 Minutes post CAC | 0.3 (0.6) | 0.6 (0.9) | 0.3 (0.5)
  15 Minutes post-dose: 20 Minutes post CAC | 0.2 (0.6) | 0.6 (1.0) | 0.4 (0.7)
  8 Hours post-dose: 7 Minutes post CAC | 0.0 (0.0) | 0.4 (0.7) | 0.1 (0.3)
  8 Hours post-dose: 15 Minutes post CAC | 0.1 (0.5) | 0.7 (0.9) | 0.2 (0.5)
  8 Hours post-dose: 20 Minutes post CAC | 0.3 (0.9) | 0.7 (1.1) | 0.3 (0.6)
  16 Hours post-dose: 7 Minutes post CAC | 0.2 (0.5) | 0.2 (0.5) | 0.1 (0.4)
  16 Hours post-dose: 15 Minutes post CAC | 0.3 (0.6) | 0.7 (1.0) | 0.4 (0.8)
  16 Hours post-dose: 20 Minutes post CAC | 0.3 (0.5) | 0.7 (1.0) | 0.6 (0.8)

10. Secondary Outcome: Nasal Congestion
Description: Nasal Congestion score: 0 = None-Breathes freely; 1.0 = Mild-Breathes with difficulty; 2.0 = Moderate-One nostril partially blocked; 3.0 = Moderate/Severe-Both nostrils partially blocked or one nostril completely blocked and the other nostril partially blocked; 4.0 = Severe-Both nostrils completely blocked
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.2 (0.5) | 0.6 (0.9) | 0.3 (0.5)
  15 Minutes post-dose: 15 Minutes post CAC | 0.3 (0.6) | 0.6 (0.9) | 0.3 (0.6)
  15 Minutes post-dose: 20 Minutes post CAC | 0.3 (0.6) | 0.6 (0.8) | 0.4 (0.7)
  8 Hours post-dose: 7 Minutes post CAC | 0.4 (0.8) | 0.6 (0.9) | 0.3 (0.7)
  8 Hours post-dose: 15 Minutes post CAC | 0.4 (0.8) | 0.8 (1.0) | 0.4 (0.9)
  8 Hours post-dose: 20 Minutes post CAC | 0.4 (0.8) | 0.8 (1.0) | 0.5 (0.9)
  16 Hours post-dose: 7 Minutes post CAC | 0.6 (0.9) | 0.7 (0.9) | 0.5 (0.7)
  16 Hours post-dose: 15 Minutes post CAC | 0.7 (0.9) | 0.8 (1.0) | 0.6 (0.8)
  16 Hours post-dose: 20 Minutes post CAC | 0.7 (0.9) | 0.7 (0.9) | 0.6 (0.8)

11. Secondary Outcome: Total Non-Ocular Composite Symptom
Description: Total Non-Ocular Composite Symptom score (Composite of Rhinorrhea, Nasal Pruritus, Ear or Palate Pruritus, and Nasal Congestion): 0 = None; 1.0 = Mild; 2.0 = Moderate; 3.0 = Moderate/Severe; 4.0 = Severe
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Units on a scale
  15 Minutes post-dose: 7 Minutes post CAC | 0.6 (1.2) | 2.2 (2.7) | 0.7 (1.2)
  15 Minutes post-dose: 15 Minutes post CAC | 1.0 (1.9) | 2.7 (3.0) | 1.1 (1.7)
  15 Minutes post-dose: 20 Minutes post CAC | 1.1 (1.8) | 2.4 (3.1) | 1.4 (2.1)
  8 Hours post-dose: 7 Minutes post CAC | 0.7 (1.5) | 2.3 (2.6) | 0.9 (1.5)
  8 Hours post-dose: 15 Minutes post CAC | 1.0 (1.7) | 3.3 (3.2) | 1.4 (2.4)
  8 Hours post-dose: 20 Minutes post CAC | 1.2 (1.9) | 3.0 (3.3) | 1.6 (2.7)
  16 Hours post-dose: 7 Minutes post CAC | 1.7 (2.1) | 2.4 (2.9) | 1.6 (1.8)
  16 Hours post-dose: 15 Minutes post CAC | 2.0 (2.3) | 3.5 (3.6) | 2.1 (2.1)
  16 Hours post-dose: 20 Minutes post CAC | 1.9 (2.3) | 3.2 (3.5) | 2.4 (2.2)

12. Secondary Outcome: Tearing
Description: Percent of Eyes with Tearing as measured 7, 15 & 20 minutes post-CAC. Scored as absent or present
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Number; unit: Percent of Eyes with Tearing Present
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Percent of Eyes with Tearing Present
  15 Minutes post-dose: 7 Minutes post CAC | 5.8 | 32.6 | 0.0
  15 Minutes post-dose: 15 Minutes post CAC | 5.8 | 23.3 | 6.8
  15 Minutes post-dose: 20 Minutes post CAC | 3.5 | 20.9 | 10.2
  8 Hours post-dose: 7 Minutes post CAC | 14.0 | 31.4 | 8.0
  8 Hours post-dose: 15 Minutes post CAC | 10.5 | 29.1 | 13.6
  8 Hours post-dose: 20 Minutes post CAC | 11.6 | 22.1 | 13.6
  16 Hours post-dose: 7 Minutes post CAC | 24.4 | 24.4 | 17.0
  16 Hours post-dose: 15 Minutes post CAC | 9.3 | 25.6 | 13.6
  16 Hours post-dose: 20 Minutes post CAC | 7.0 | 17.4 | 14.8

13. Secondary Outcome: Ocular Mucus Discharge
Description: Percent of Eyes with Ocular Mucus Discharge as measured 7, 15 & 20 minutes post-CAC.
  Scored as absent or present
Time Frame: 15 Minutes, 8 Hours & 16 Hours post-dose from Conjunctival Allergen Challenge (CAC) Model
Measure: Number; unit: Percent of Eyes with OMD Present
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Number analyzed (Participants) | 43 | 43 | 44
Percent of Eyes with OMD Present
  15 Minutes post-dose: 7 Minutes post CAC | 2.3 | 0.0 | 0.0
  15 Minutes post-dose: 15 Minutes post CAC | 1.2 | 1.2 | 0.0
  15 Minutes post-dose: 20 Minutes post CAC | 1.2 | 1.2 | 0.0
  8 Hours post-dose: 7 Minutes post CAC | 1.2 | 8.1 | 0.0
  8 Hours post-dose: 15 Minutes post CAC | 3.5 | 10.5 | 0.0
  8 Hours post-dose: 20 Minutes post CAC | 4.7 | 7.0 | 1.1
  16 Hours post-dose: 7 Minutes post CAC | 1.2 | 0.0 | 0.0
  16 Hours post-dose: 15 Minutes post CAC | 0.0 | 0.0 | 0.0
  16 Hours post-dose: 20 Minutes post CAC | 0.0 | 0.0 | 2.3

ADVERSE EVENTS:
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo | Bepotastine Besilate Ophthalmic Solution 1.0%
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 3/43 | 3/43 | 5/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% (N=43) | Placebo (N=43) | Bepotastine Besilate Ophthalmic Solution 1.0% (N=44)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement is between contract research organization and third parties on behalf of ISTA Pharmaceuticals, Inc.